CLINICAL TRIAL: NCT05130099
Title: A Complex Intervention for a Complex Symptom - a Randomized Controlled Trial in Chronically Fatigued Lymphoma Survivors
Brief Title: A Complex Intervention for Chronically Fatigued Lymphoma Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian School of Sport Sciences (Other); UiT The Arctic University of Norway (Other); Norwegian University of Science and Technology (Other); Diakonhjemmet Hospital (Other); University of Alberta (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Lene Thorsen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: #153665
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Chronic Fatigue Syndrome
Keywords: lymphoma; cancer survivorship; physical activity; nutrition; patient education; cognitive behavioral program
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Lymphoma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary complex intervention (Experimental)
  Interventions: Other: Interdisciplinary complex intervention
- Usual care (No Intervention): Six months after the intervention period (T3), the participants randomized to usual care will be offered a modified version of the intervention in line with their personally expressed needs.

INTERVENTIONS:
Other: Interdisciplinary complex intervention — The interdisciplinary complex intervention lasts 12 weeks and includes the 4 following components;
  Patient-education: a 2-hours group-based digital session, including information about fatigue, training theory, psychological strategies and nutrition, all in relation to chronic fatigue (CF).
  Physical exercise program: two weekly sessions with aerobic exercise and resistance training. The participants are instructed to do the same program in the unsupervised sessions as in the supervised sessions. After the first 12 weeks exercise period, the participant and the physiotherapist makes an individually tailored plan for exercise and follow-up the next 12 weeks.
  Cognitive behavioral program: 6 group-based online sessions lead by two psychologists, based on elements from cognitive behavioral therapy to reduce and/or manage CF. Each session lasts for 135 minutes.
  Nutritional counselling: 3 individual sessions by a clinical dietitian. Each session lasts for 30-60 minutes.
  Arms: Interdisciplinary complex intervention

SUMMARY:
The present study is a randomized controlled trial (RCT) with an overall objective to examine the effect of an interdisciplinary complex intervention on the level of fatigue in lymphoma survivors with chronic fatigue. Secondary aims are to examine the effects of the intervention on daily functioning, work status/ability, physical fitness and QoL among the survivors, on QoL of their relatives and on the societal costs.The intervention will last for 12+12 weeks and include four components; patient education, supervised physical exercise, cognitive behavioral program and nutritional counselling. Outcomes will be assessed at baseline,post-intervention (12 weeks after baseline) and at 3-month, 6-month, 12-month and 24-month follow-up after completed intervention.

DETAILED DESCRIPTION:
Chronic fatigue (CF) is a subjective experience of substantial lack of energy, exhaustion and cognitive difficulties lasting for six months or longer. CF is one of the most common and distressing late effects after cancer, affecting 15-35 % of survivors, often for years beyond treatment. Despite the high prevalence and the huge negative consequences of CF on daily functioning and QoL and the economic and societal costs, effective treatment of CF and standardized follow-up care are currently lacking.

Today, there is no curative treatment of CF. However, several modifiable behavioral factors including emotional distress, physical inactivity, sleep disturbances and unhealthy diets are found to be associated with CF. So far, most of the interventions aiming to reduce fatigue during and shortly after cancer treatment have targeted only one of these factors at a time, with small to moderate effect sizes. No prior study has examined if CF in cancer survivors is better treated by a complex intervention targeting combinations of these factors, an approach which seems logical due to the complexity of the symptom.

The project is a two-armed RCT in which chronically fatigued lymphoma survivors are randomized to an interdisciplinary complex intervention or to usual care. Eligible participants will receive written information about the study by mail. Survivors who perceive themselves as having physical and mental fatigue, and who are willing to participate, will be asked to fill out and return the Chalder Fatigue Questionnaire (FQ) to the study coordinator. Those who have chronic fatigue as measured by the FQ will be invited to a medical screening by an oncologist in the project group, for evaluation of inclusion.

The interdisciplinary complex intervention will last for 12 + 12 weeks and include four components; patient education, physical exercise (and follow-up), cognitive behavioral program and nutritional counselling, organized in a systematic way, i.e. a standardized patient care pathway.

All outcomes will be assessed in all participants at four points; pre-intervention (baseline) (T0), post-intervention (12 weeks after baseline) (T1) and at 3-month (T2) and 6-month (T3) after T1. Moreover, selected patient reported outcomes will be assessed in all participants at 12-month (T4) and 24-month (T5) after T1.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of Hodgkin and aggressive non-Hodgkin lymphoma
* Not indolent non-Hodgkin lymphoma
* Not CNS lymphoma at diagnosis
* Not second cancer
* Not ongoing cancer treatment
* Chronic fatigue measured by Chalder Fatigue Questionnaire
* Diagnosed 2010-2020
* Received treatment with curative intent
* 18 - 70 years old at inclusion
* > 2 years since last treatment
* Able to understand the Norwegian language
* Participation approval from oncologist in the project group

Exclusion Criteria:

* Persisting fatigue > 1 year before the cancer diagnosis
* Somatic/physical conditions (i.e. severe heart failure/disease, lung disease, use of wheelchair /crutches)
* Psychiatric or mental disorders (i.e. dementia, severe depression, schizophrenia)
* Use of stimulants for ADHD
* Substance abuse disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in change in fatigue levels (physical-, mental- and total fatigue) between intervention and control group, assessed by the Chalder Fatigue Questionnaire | From baseline (T0) to 12 weeks (T1)
  The Fatigue Questionnaire consists of 11 questions, distributed on a physical fatigue scale (7 items) and mental fatigue scale (4 items) Each item is scored from 0 to 3. This provides a physical fatigue score from 0 to 21, mental fatigue score from 0 to 12, and total score from 0 to 33. Higher score implies more fatigue.

SECONDARY OUTCOMES:
Difference in change in fatigue levels between groups assessed by Chalder Fatigue Questionnaire | From baseline (T0) to 24 weeks (T2)
  The Fatigue Questionnaire consists of 11 questions, distributed on a physical fatigue scale (7 items) and mental fatigue scale (4 items) Each item is scored from 0 to 3, providing a total score from 0 to 33. Higher score implies more fatigue.
Difference in change in fatigue levels between groups assessed by Chalder Fatigue Questionnaire | From baseline (T0) to 36 weeks (T3)
  The Fatigue Questionnaire consists of 11 questions, distributed on a physical fatigue scale (7 items) and mental fatigue scale (4 items) Each item is scored from 0 to 3, providing a total score from 0 to 33. Higher score implies more fatigue.
Change in fatigue levels among all participants assessed by Chalder Fatigue Questionnaire | From post-intervention (T1) to 12-month follow-up (T4)
  The Fatigue Questionnaire consists of 11 questions, distributed on a physical fatigue scale (7 items) and mental fatigue scale (4 items) Each item is scored from 0 to 3, providing a total score from 0 to 33. Higher score implies more fatigue.
Change in fatigue levels among all participants assessed by Chalder Fatigue Questionnaire | From post-intervention (T1) to 24-month follow-up (T5)
  The Fatigue Questionnaire consists of 11 questions, distributed on a physical fatigue scale (7 items) and mental fatigue scale (4 items) Each item is scored from 0 to 3, providing a total score from 0 to 33. Higher score implies more fatigue.
Difference in change in daily functioning between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 12 weeks (T1)
  The questionnaire includes five functioning scales (physical, role, cognitive, emotional and social).All of the scales range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning.
Difference in change in daily functioning between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 24 weeks (T2)
  The questionnaire includes five functioning scales (physical, role, cognitive, emotional and social).All of the scales range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning.
Difference in change in daily functioning between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 36 weeks (T3)
  The questionnaire includes five functioning scales (physical, role, cognitive, emotional and social).All of the scales range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning.
Change in daily functioning among all participants assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From post-intervention (T1) to 12-month follow-up (T4)
  The questionnaire includes five functioning scales (physical, role, cognitive, emotional and social).All of the scales range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning.
Change in daily functioning among all participants assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From post-intervention (T1) to 24-month follow-up (T5)
  The questionnaire includes five functioning scales (physical, role, cognitive, emotional and social).All of the scales range in score from 0 to 100.
  A high score for a functional scale represents a high / healthy level of functioning.
Difference in change in global quality of life between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 12 weeks (T1)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in global quality of life between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 24 weeks (T2)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in global quality of life between groups assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 36 weeks (T3)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Change in global quality of life among all participants assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From post-intervention (T1) to 12-month follow-up (T4)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Change in global quality of life among all participants assessed by European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From post-intervention (T1) to 24-month follow-up (T5)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in work status between groups assessed by questions from the HUNT4-study | From baseline (T0) to 12 weeks (T1)
  Participants are asked to report their current work status
Difference in change in work status between groups assessed by questions from the HUNT4-study | From baseline (T0) to 24 weeks (T2)
  Participants are asked to report their current work status
Difference in change in work status between groups assessed by questions from the HUNT4-study | From baseline (T0) to 36 weeks (T3)
  Participants are asked to report their current work status
Change in work status in both groups assessed by questions from the HUNT4-study | From post-intervention (T1) to 12 months follow-up (T4)
  Participants are asked to report their current work status
Change in work status in both groups assessed by questions from the HUNT4-study | From post-intervention (T1) to 24 months follow-up (T5)
  Participants are asked to report their current work status
Difference in change in work ability between groups assessed by the Work Ability Index scale | From baseline (T0) to 12 weeks (T1)
  Current work ability is rated compared with the lifetime best on a scale from 0 to 10. Higher score implies higher work ability.
Difference in change in work ability between groups assessed by the Work Ability Index scale | From baseline (T0) to 24 weeks (T2)
  Current work ability is rated compared with the lifetime best on a scale from 0 to 10. Higher score implies higher work ability.
Difference in change in work ability between groups assessed by the Work Ability Index scale | From baseline (T0) to 36 weeks (T3)
  Current work ability is rated compared with the lifetime best on a scale from 0 to 10. Higher score implies higher work ability.
Change in work ability in both groups assessed by the Work Ability Index scale | From post-intervention (T1) to 12 months follow-up (T4)
  Current work ability is rated compared with the lifetime best on a scale from 0 to 10. Higher score implies higher work ability.
Change in work ability in both groups assessed by the Work Ability Index scale | From post-intervention (T1) to 24 months follow-up (T5)
  Current work ability is rated compared with the lifetime best on a scale from 0 to 10. Higher score implies higher work ability.
Difference in change in work ability between groups assessed by the Work Ability Index: physical demands of the job | From baseline (T0) to 12 weeks (T1)
  Assessed by rating work ability in relation to the physical demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in work ability between groups assessed by the Work Ability Index: physical demands of the job | From baseline (T0) to 24 weeks (T2)
  Assessed by rating work ability in relation to the physical demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in work ability between groups assessed by the Work Ability Index: physical demands of the job | From baseline (T0) to 36 weeks (T3)
  Assessed by rating work ability in relation to the physical demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Change in work ability in both groups assessed by the Work Ability Index: physical demands of the job | From post-intervention (T1) to 12 months follow-up (T4)
  Assessed by rating work ability in relation to the physical demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Change in work ability in both groups assessed by the Work Ability Index: physical demands of the job | From post-intervention (T1) to 24 months follow-up (T5)
  Assessed by rating work ability in relation to the physical demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in work ability between groups assessed by the Work Ability Index: psychological demands of the job | From baseline (T0) to 12 weeks (T1)
  Assessed by rating work ability in relation to the psychological demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in work ability between groups assessed by the Work Ability Index: psychological demands of the job | From baseline (T0) to 24 weeks (T2)
  Assessed by rating work ability in relation to the psychological demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in work ability between groups assessed by the Work Ability Index: psychological demands of the job | From baseline (T0) to 36 weeks (T3)
  Assessed by rating work ability in relation to the psychological demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Change in work ability in both groups assessed by the Work Ability Index: psychological demands of the job | From post-intervention (T1) to 12 months follow-up (T4)
  Assessed by rating work ability in relation to the psychological demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Change in work ability in both groups assessed by the Work Ability Index: psychological demands of the job | From post-intervention (T1) to 24 months follow-up (T5)
  Assessed by rating work ability in relation to the psychological demands of the job, by the following response alternatives: very good, rather good, moderate, rather poor or very poor
Difference in change in cardiorespiratory fitness between groups assessed by cardio-pulmonary exercise testing (CPET) | From baseline (T0) to 12 weeks (T1)
  Peak oxygen uptake (VO2peak) is measured
Difference in change in cardiorespiratory fitness between groups assessed by cardio-pulmonary exercise testing (CPET) | From baseline (T0) to 24 weeks (T2)
  Peak oxygen uptake (VO2peak) is measured
Difference in change in cardiorespiratory fitness between groups assessed by cardio-pulmonary exercise testing (CPET) | From baseline (T0) to 36 weeks (T3)
  Peak oxygen uptake (VO2peak) is measured
Difference in change in cardiorespiratory fitness between groups assessed by a treadmill test | From baseline (T0) to 12 weeks (T1)
  In cases where participants do not have the opportunity to travel for physical fitness tests, cardiorespiratory fitness will be assessed by an indirect treadmill test (modified Balke protocol) at their local physiotherapist. Time to exhaustion will be used as an indicator of cardiorespiratory fitness.
Difference in change in cardiorespiratory fitness between groups assessed by a treadmill test | From baseline (T0) to 24 weeks (T2)
  In cases where participants do not have the opportunity to travel for physical fitness tests, cardiorespiratory fitness will be assessed by an indirect treadmill test (modified Balke protocol) at their local physiotherapist. Time to exhaustion will be used as an indicator of cardiorespiratory fitness.
Difference in change in cardiorespiratory fitness between groups assessed by a treadmill test | From baseline (T0) to 36 weeks (T3)
  In cases where participants do not have the opportunity to travel for physical fitness tests, cardiorespiratory fitness will be assessed by an indirect treadmill test (modified Balke protocol) at their local physiotherapist. Time to exhaustion will be used as an indicator of cardiorespiratory fitness.
Difference in change in lower body muscle strength between groups assessed by leg press | From baseline (T0) to 12 weeks (T1)
  The one-repetition maximum (1RM) test (the maximal workload that can be lifted once)) in leg press.
Difference in change in lower body muscle strength between groups assessed by leg press | From baseline (T0) to 24 weeks (T2)
  The one-repetition maximum (1RM) test (the maximal workload that can be lifted once)) in leg press.
Difference in change in lower body muscle strength between groups assessed by leg press | From baseline (T0) to 36 weeks (T3)
  The one-repetition maximum (1RM) test (the maximal workload that can be lifted once)) in leg press.
Difference in change in lower body muscle strength between groups assessed by push-ups | From baseline (T0) to 12 weeks (T1)
  The maximum number of push-ups that can be performed in one set
Difference in change in upper body muscle strength between groups assessed by push-ups | From baseline (T0) to 24 weeks (T2)
  The maximum number of push-ups that can be performed in one set
Difference in change in upper body muscle strength between groups assessed by push-ups | From baseline (T0) to 36 weeks (T3)
  The maximum number of push-ups that can be performed in one set
Difference in change in level of depressive symptoms between groups assessed by the Patient Health Questionnaire-9 | From baseline (T0) to 12 weeks (T1)
  Each of the 9 items is scored from 0-3, providing a total score from 0 to 27. A higher score implies higher level of depressive symptoms.
Difference in change in level of depressive symptoms between groups assessed by the Patient Health Questionnaire-9 | From baseline (T0) to 24 weeks (T2)
  Each of the 9 items is scored from 0-3, providing a total score from 0 to 27. A higher score implies higher level of depressive symptoms.
Difference in change in level of depressive symptoms between groups assessed by the Patient Health Questionnaire-9 | From baseline (T0) to 36 weeks (T3)
  Each of the 9 items is scored from 0-3, providing a total score from 0 to 27. A higher score implies higher level of depressive symptoms.
Change in level of depressive symptoms among all participants assessed by the Patient Health Questionnaire-9 | From post-intervention (T1) to 12-month follow-up (T4)
  Each of the 9 items is scored from 0-3, providing a total score from 0 to 27. A higher score implies higher level of depressive symptoms.
Change in level of depressive symptoms among all participants assessed by the Patient Health Questionnaire-9 | From post-intervention (T1) to 24-month follow-up (T5)
  Each of the 9 items is scored from 0-3, providing a total score from 0 to 27. A higher score implies higher level of depressive symptoms.
Difference in change in level of anxiety symptoms between groups assessed by the General Anxiety Disorder 7-items (GAD7). | From baseline (T0) to 12 weeks (T1)
  Each of the 7 items is scored from 0-3, providing a total score from 0-21. A higher score implies higher level of anxiety symptoms.
Difference in change in level of anxiety symptoms between groups assessed by the General Anxiety Disorder 7-items (GAD7). | From baseline (T0) to 24 weeks (T2)
  Each item is scored from 0-3, providing a total score from 0-21. A higher score implies higher level of anxiety symptoms.
Difference in change in level of anxiety symptoms between groups assessed by the General Anxiety Disorder 7-items (GAD7). | From baseline (T0) to 36 weeks (T3)
  Each of the 7 items is scored from 0-3, providing a total score from 0-21. A higher score implies higher level of anxiety symptoms.
Change in level of anxiety symptoms in all participants assessed by the General Anxiety Disorder 7-items (GAD7). | From baseline (T0) to 12 months follow-up weeks (T4)
  Each of the 7 items is scored from 0-3, providing a total score from 0-21. A higher score implies higher level of anxiety symptoms.
Change in level of anxiety symptoms in all participants assessed by the General Anxiety Disorder 7-items (GAD7). | From baseline (T0) to 24 months follow-up weeks (T5)
  Each of the 7 items is scored from 0-3, providing a total score from 0-21. A higher score implies higher level of anxiety symptoms.
Difference in change in sense of exercise competence between groups assessed by the Perceived Competence Scale. | From baseline (T0) to 12 weeks (T1)
  The scale consists of 4 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 0 to 7 is calculated based on the mean score of the items, with increasing score implying higher exercise competence.
Difference in change in sense of exercise competence between groups assessed by the Perceived Competence Scale. | From baseline (T0) to 24 weeks (T2)
  The scale consists of 4 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 0 to 7 is calculated based on the mean score of the items, with increasing score implying higher exercise competence.
Difference in change in sense of exercise competence between groups assessed by the Perceived Competence Scale. | From baseline (T0) to 36 weeks (T3)
  The scale consists of 4 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 0 to 7 is calculated based on the mean score of the items, with increasing score implying higher exercise competence.
Change in sense of exercise competence in both groups assessed by the Perceived Competence Scale. | From post-intervention (T1) to 12 months follow-up (T4)
  The scale consists of 4 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 0 to 7 is calculated based on the mean score of the items, with increasing score implying higher exercise competence.
Change in sense of exercise competence in both groups assessed by the Perceived Competence Scale. | From post-intervention (T1) to 24 months follow-up (T5)
  The scale consists of 4 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 0 to 7 is calculated based on the mean score of the items, with increasing score implying higher exercise competence.
Difference in change in satisfaction with life between groups assessed by the Satisfaction With Life Scale. | From baseline (T0) to 12 weeks (T1)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher satisfaction with life.
Difference in change in satisfaction with life between groups assessed by the Satisfaction With Life Scale. | From baseline (T0) to 24 weeks (T2)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher satisfaction with life.
Difference in change in satisfaction with life between groups assessed by the Satisfaction With Life Scale. | From baseline (T0) to 36 weeks (T3)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher satisfaction with life.
Difference in change in sense of vitality between groups assessed by the Subjective Vitality Scale | From baseline (T0) to 12 weeks (T1)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher sense of vitality.
Difference in change in sense of vitality between groups assessed by the Subjective Vitality Scale | From baseline (T0) to 24 weeks (T2)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher sense of vitality.
Difference in change in sense of vitality between groups assessed by the Subjective Vitality Scale | From baseline (T0) to 36 weeks (T3)
  The scale consists of 5 items, each scored from 1 (totally disagree) to 7 (totally agree). A sum score from 5 to 35 is calculated, with increasing score implying higher sense of vitality.
Difference in change in adherence to the Norwegian food-based dietary guidelines between groups assessed by DIGIKOST-FFQ | From baseline (T0) to 12 weeks (T1)
  DIGIKOST-FFQ is a food frequency questionnaire aiming to benchmark against the Norwegian food-based dietary guidelines.
Difference in change in adherence to the Norwegian food-based dietary guidelines assessed by DIGIKOST-FFQ | From baseline (T0) to 24 weeks (T2)
  DIGIKOST-FFQ is a food frequency questionnaire aiming to benchmark against the Norwegian food-based dietary guidelines.
Difference in change in adherence to the Norwegian food-based dietary guidelines assessed by DIGIKOST-FFQ | From baseline (T0) to 36 weeks (T3)
  DIGIKOST-FFQ is a food frequency questionnaire aiming to benchmark against the Norwegian food-based dietary guidelines.
Difference in change in general health between groups measured by European Quality of Life Five-Dimension Scale Questionnaire (EQ-5D) | From baseline (T0) to 12 weeks (T1)
  EQ-5D consists of five dimensions (mobility, self-care, usual activities, pain & discomfort, anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Difference in change in general health between groups measured by European Quality of Life Five-Dimension Scale Questionnaire (EQ-5D) | From baseline (T0) to 24 weeks (T2)
  EQ-5D consists of five dimensions (mobility, self-care, usual activities, pain & discomfort, anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Difference in change in general health between groups measured by European Quality of Life Five-Dimension Scale Questionnaire (EQ-5D) | From baseline (T0) to 36 weeks (T3)
  EQ-5D consists of five dimensions (mobility, self-care, usual activities, pain & discomfort, anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
Difference in change in quality of life among the relatives between groups measured by Research and Development 36-term Short Form Health Survey (RAND SF-36) | From baseline (T0) to 12 weeks (T1)
  RAND-36 comprises 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales.All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Difference in change in quality of life among the relatives between groups measured by Research and Development 36-term Short Form Health Survey (RAND SF-36) | From baseline (T0) to 24 weeks (T2)
  RAND-36 comprises 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales.All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Difference in change in quality of life among the relatives between groups measured by Research and Development 36-term Short Form Health Survey (RAND SF-36) | From baseline (T0) to 36 weeks (T3)
  RAND-36 comprises 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales.All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible.
Difference in change in quality of life among the relatives between groups measured by the global health status / QoL scale from the European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 12 weeks (T1)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in quality of life among the relatives between groups measured by the global health status / QoL scale from the European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 24 weeks (T2)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in quality of life among the relatives between groups measured by the global health status / QoL scale from the European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 36 weeks (T2)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Difference in change in quality of life among the relatives between groups measured by the global health status / QoL scale from the European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). | From baseline (T0) to 36 weeks (T3)
  The questionnaire includes a global health status / quality of life (QoL) scale, which range in score from 0 to 100. A high score for the global health status / QoL represents a high QoL.
Cost-effectiveness of the intervention, calculated based on measurements of health-related QoL and resource use (costs related to the intervention). | From baseline (0) to 36 weeks (T3)
  Combining information about health-related QoL will give quality-adjusted life-years, while valuation of resource use using standard principles of health economic evaluation will provide estimates of costs
Perceived benefits of the intervention components assessed by questions used in and modified from the PasOpp study from the Directorate of Health in Norway | At 12- and 24-month follow-up
  Questions assessing benefits of the intervention
Use of information, experiences, strategies and advices learned in the intervention program assessed by self-made questions | At 12- and 24-month follow-up
  Questions assessing daily use of information, strategies and advices learned in the intervention program

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Bohn SH, Reinertsen KV, Kiserud CE, Loge JH, Fossa A, Skaali T, Blomhoff R, Oldervoll LM, Courneya KS, Raastad T, Nilsen TS, Wisloff T, Lie HC, Berge T, Edvardsen E, Fagerli UM, Fjerstad E, Gjerset GM, Haavik I, Henriksen HB, Rutkovskiy A, Sandberg G, Seland M, Slott M, Tjessem KH, Viktil L, Thorsen L. Effects of a Multidisciplinary Intervention on Fatigue in Lymphoma Survivors With Chronic Fatigue: Protocol for a Randomized Controlled Trial (REFUEL). JMIR Res Protoc. 2025 Aug 29;14:e69336. doi: 10.2196/69336. PMID 40882189